CLINICAL TRIAL: NCT00675831
Title: Infusion of Donor Lymphocytes Depleted of CD25+ Regulatory T-cells in Patients With Relapsed Hematologic Malignancies After Matched Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Infusion of Donor Lymphocytes Depleted of CD25+ Regulatory T-cells in Patients With Relapsed Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Principal Investigator, John Koreth, MD, MBBS, DPhil, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-193
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Hematologic Malignancies
Keywords: CD25+; Tregs; DLI; Donor lymphocyte infusion
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD25+ Treg depleted DLI dose schema (Experimental): Patients will receive a defined dose of CD25+ Treg depleted DLI. 5 patients will be enrolled, initially at dose level B, and subsequent cohorts will be dose adjusted per the CD3+ dose escalation/de-escalation schema:
  * Dose level -C: 3x10^7 (CD3+Dose (#cells/kg*))
  * Dose level -B: 1x10^7 (CD3+Dose (#cells/kg*))
  * Dose level -A: 1x10^6 (CD3+Dose (#cells/kg*)) *Recipient's body weight in Kg
  Interventions: Device: CliniMACS CD25 Reagent Device

INTERVENTIONS:
Device: CliniMACS CD25 Reagent Device — Used to engineer CD25+ depleted donor lymphocytes which will be infused intravenously over 5-10 minutes

SUMMARY:
The purpose of this research study is to evaluate the safety and efficacy of cell depletion in a donor lymphocyte infusion (DLI) product with the use of the CliniMACS machine. Previously, patients with hematologic malignancies who have relapsed after transplant have been given infusions of donor white blood cells calsed donor lymphocyte infusion (DLI) as a way to boost their immune function and fight cancer. Information from other research studies suggests that lowering the number of a certain type of white blood cell called CD25+ Tregs in the DLI may allow for a greater effect. In this research study, we are looking for the appropriate dose of DLI depleted of the CD25+ Treg white blood cells that can be given safely.

DETAILED DESCRIPTION:
* The original marrow/stem cell donor will undergo one or two white blood cell collection procedures called leukopheresis. The cells collected from the first leukopheresis will be sent to the laboratory where the amount of white blood cells collected will be measured. If the number of cells collected at the first leukopheresis is not enough, the donor will have a second leukopheresis procedure.
* Once enough lymphocytes are collected from the donor, the CliniMACS CD25 Reagent System device will reduce the number of CD25+ Tregs. The CD25+ depleted donor lymphocytes will then be infused to the participant intravenously. Participants will be observed for about one hour after the infusion.
* One, two, four and eight weeks after the DLI, participants will return to the clinic for follow-up visits. At each visit a physical exam, questions about the participants general health, and blood tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies that have relapsed after HLA-A, -B, -C, and-DRBI matched allogeneic hematopoietic stem cell transplantation
* At least 2 months following hematopoietic stem cell transplantation
* Off any systemic immunosuppressive medication for treatment or prevention of GVHD, for a minimum of 2 weeks prior to study entry
* Recipient with donor chimerism of 20% or greater within 6 weeks prior to DLI
* Patient with less than 50% bone marrow involvement (% cellularity) and less than 5cm lymph nodes, in the 6 weeks prior to DLI
* 18 years of age or older
* ECOG Performance Status score 0-2
* Prior stem cell donor is medically fit to undergo leukapheresis procedure

Exclusion Criteria:

* Relapsed CML in chronic phase
* Prior donor lymphocyte infusion or other immunotherapy treatment within 8 weeks prior to enrollment
* Chemotherapy within 4 weeks prior to enrollment
* Clinically significant and active autoimmune disease in donor or patient. This is defined as autoimmune disease resulting in organ dysfunction and/or requiring systemic therapy
* Evidence of active acute or chronic GVHD
* Uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of using the ClinMACS CD25 Reagent device to engineer a DLI product outlined in the protocol | 3 years
To determine the safety of CD25+ Treg depleted DLI in this patient population. | 3 years

SECONDARY OUTCOMES:
To assess clinical response after infusions of CD25+ Treg depleted donor lymphocytes | 3 years
To assess the immunologic impact of infusions of CD25+ Treg depleted donor lymphocytes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MBBS, DPhil, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nikiforow S, Kim HT, Daley H, Reynolds C, Jones KT, Armand P, Ho VT, Alyea EP 3rd, Cutler CS, Ritz J, Antin JH, Soiffer RJ, Koreth J. A phase I study of CD25/regulatory T-cell-depleted donor lymphocyte infusion for relapse after allogeneic stem cell transplantation. Haematologica. 2016 Oct;101(10):1251-1259. doi: 10.3324/haematol.2015.141176. Epub 2016 Jun 27. PMID 27354021